CLINICAL TRIAL: NCT04404231
Title: Treatment of Intrapartum Depression Using Non-invasive Photobiomodulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Maurice-Andre Recanati, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 20-05-2295
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Depression; Pregnancy Related; Intrapartum Depression
Keywords: photobiomodulation; intrapartum depression; phototherapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and the investigator are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No infrared light therapy (Sham Comparator): This arm does not receive any phototherapy
  Interventions: Other: No Infrared treatment
- 810 nm (Active Comparator): Many clinical studies have used 810nm twice a week for 4 weeks. This is the standard.
  Interventions: Radiation: Delivery of infrared light to the head
- 945nm (Experimental): This wavelength has been chosen as a comparison to 810, to see if it works better.
  Interventions: Radiation: Delivery of infrared light to the head
- random frequency (Experimental): A wavelength between 650-1100nm which is picked at random
  Interventions: Radiation: Delivery of infrared light to the head

INTERVENTIONS:
Radiation: Delivery of infrared light to the head — Building upon the experience gathered from previous depression clinical trials, we will treat twice weekly for a total of 4-week duration consisting of 8 sessions. Each treatment will last 20 min and areas irradiated will include frontal and temporal areas bilaterally. Irradiance of 250 mW/cm2 with a fluence of 60 J/cm2.
  Arms: 810 nm; 945nm; random frequency
Other: No Infrared treatment — This is sham treatment. No light is actually given.
  Arms: No infrared light therapy

SUMMARY:
Depression during pregnancy can cause fetal and maternal problems such as growth restriction, preterm labor, low birthweight, poor compliance and suicide. Since antidepressant medications have the potential to harm the baby, but since treatment of intrapartum depression is essential to maternal and fetal wellbeing, a non-pharmacological approach would be ideal. This project seeks to apply infrared light noninvasively to depressed patients during pregnancy in order to treat depressive symptoms through alteration of mitochondrial function and modulation of neural cell receptors.

DETAILED DESCRIPTION:
Depression is common in pregnancy and affects about 70% of women and, for many women, pregnancy can lead to the first episode of major depression. Complications of intrapartum depression include intrauterine growth restriction, preterm labor, low birthweight, gestational diabetes, preeclampsia, decreased prenatal follow-up and suicide. For this reason, the standard of care has been to screen for depression during pregnancy and treat this illness, reducing maternal and fetal morbidity. Unfortunately, many first-line pharmacological approaches, such as serotonin reuptake inhibitors, may cause fetal malformations, persistent pulmonary hypertension and withdrawal syndrome. Thus, a non-pharmacological approach, without risk of fetal complications, would be ideal. The investigators propose a photobiomodulation based approach that uses non-ionizing near-infrared light (IRL) to upregulate mitochondrial function (through modulation of cytochrome c oxidase activity), which in-turn increase neurosteroid production and modulates GABAA receptor activity, thus alleviating depression. The investigators will perform a pilot study using IRL for the treatment of intrapartum depression. While other trials have shown success using IRL for depression in non-pregnant patients, this will confirm that photobiomodulation can modulate mitochondrial function and mitigate depressive symptoms compared to untreated controls in pregnancy by using real-time app-based depression scoring system and neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Viable intrauterine pregnancy <16 weeks, PHQ-9 or Edinburg Score>10.

Exclusion Criteria:

* pregnancy > 20 weeks
* history of seizures
* history of migraines
* history of multiple sclerosis
* prior traumatic brain injury
* prior history of preeclampsia/toxemia
* elevated blood pressure greater than 140/90
* proteinuria (as defined by urine proteins >300 mg/24 h)
* headaches
* visual changes
* right upper quadrant pain
* history of bipolar disease
* currently taking psychotropic medications (including antidepressants) and
* prior history of attempted suicide

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression score | Twice daily for the duration of the 4 week study
  Using an App based approach, patients will enter their depression score

SECONDARY OUTCOMES:
Alteration in brain metabolism | Twice. One imaging study before treatment and one at the end of the 4 weeks of treatment
  Functional MRI will be done to assess brain function and determine the effect of infrared light treatment on brain metabolics

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Medical Ceter, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Askalsky P, Iosifescu DV. Transcranial Photobiomodulation For The Management Of Depression: Current Perspectives. Neuropsychiatr Dis Treat. 2019 Nov 22;15:3255-3272. doi: 10.2147/NDT.S188906. eCollection 2019. PMID 31819453
- [Result] Cassano P, Petrie SR, Mischoulon D, Cusin C, Katnani H, Yeung A, De Taboada L, Archibald A, Bui E, Baer L, Chang T, Chen J, Pedrelli P, Fisher L, Farabaugh A, Hamblin MR, Alpert JE, Fava M, Iosifescu DV. Transcranial Photobiomodulation for the Treatment of Major Depressive Disorder. The ELATED-2 Pilot Trial. Photomed Laser Surg. 2018 Dec;36(12):634-646. doi: 10.1089/pho.2018.4490. Epub 2018 Oct 20. PMID 30346890